CLINICAL TRIAL: NCT04911179
Title: Effect of an Individualized Combined Intervention (Vivifrail-Cogn) on the Rate of Falling of Frail Older Adults at Risk of Falling Living in the Community: a Multicenter Randomized Clinical Trial.
Brief Title: Combined Exercise and Cognitive Stimulation for Falls Prevention
Acronym: Vivifrailcogn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PI20/01546
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Fall; Frailty; Cognition Disorders in Old Age; Exercise; Cognitive Change
Keywords: Fall; Frailty; Cognition Disorders in Old Age; Exercise; Cognitive Change
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined multicomponent physical exercise and cognitive stimulation (Vivfrail-Cog) (Experimental): The supervised multicomponent exercise training program (resistance, endurance, balance and flexibility) will be comprised of upper and lower body exercises tailored to the individual's functional capacity. Subjects will be encouraged at performing strength and endurance exercise at a moderate intensity. Exercise will progress in terms of intensity and difficulty upon individual adaptation.
  The cognitive intervention will include the performance of different exercises with pencil and paper in order to train different cognitive areas, especially the executive functions.
  Interventions: Other: Vivfrail-Cog combined multicomponent physical exercise and cognitive stimulation.
- Usual care (No Intervention): The usual care group will receive normal outpatient care (including the evidence-based Otago exercise program).

INTERVENTIONS:
Other: Vivfrail-Cog combined multicomponent physical exercise and cognitive stimulation. — The areas to be worked on are: Attentional system: selective attention and concentration; alternating attention / dual attention; Processing speed; perceptual organization; working memory and cognitive flexibility; comprehension, abstraction and verbal reasoning, planning, execution, and problem solving.
  Four programs have been developed stimulation different difficulty levels to adapt to the capabilities of each participant.
  Arms: Combined multicomponent physical exercise and cognitive stimulation (Vivfrail-Cog)

SUMMARY:
Randomized clinical trial of 310 older adults over 75 years old recruited from the Falls Units of Geriatric Departments in 4 three University Hospitals in Spain (Pamplona, San Sebastián, Albacete and Barcelona). Participants who met inclusion criteria will be randomized to the usual care group (Otago exercise program) or the Vivifrail-Cog Intervention (a combination of physical exercise Vivifrail program and cognitive training). The main objective of the present randomized clinical trial is to investigate the effect of the combined intervention (exercise and cognitive intervention) in frail older participants living in the community and at risk of falling. The main endpoint will be the rate of falling in the following year. Secondary endpoints include physical performance, muscle strength, cognitive performance, hospitalizations, institutionalization, depression and quality of life.

DETAILED DESCRIPTION:
Usual care: subjects randomized to the usual care group will receive an evidence-based multidisciplinary intervention tailored at reducing the fall risk (polypharmacy, environmental intervention, physical exercise). Importantly, the Otago exercise program (considered the standard physical exercise intervention) will be prescribed in this group.

Intervention group: subjects assigned to this intervention will engage in a multicomponent intervention combining an exercise program, Vivifrail (A practical guide for prescribing a Multicomponent Physical Training Program to prevent weakness and falls in people over 70, more information at www.vivifrail.com) and a cognitive training. Vivifrail exercise program combines resistance, endurance, balance and flexibility exercise tailored to the functional level of the subjects, guaranteeing an individualized approach. Exercises progress in terms of intensity and difficulty as the subject adapts to exercise. The cognitive stimulation program combines exercises to work on different cognitive functions, mainly addressing executive functions (attentional system, processing speed, perceptual organization, working memory and cognitive flexibility, verbal comprehension, abstraction and reasoning, planning, execution and problem solving ).

It lasts 12 weeks, two weekly sessions. It is divided into 4 levels in order to adapt the intervention to participant's individual capacity, and the level can be adjusted throughout the intervention.

Correct execution will be monitored by constant contact with relatives in charge of supervising the exercise program, who will be familiarized with the intervention prior to participation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years or older
* Referral to the Falls Unit
* Ability to ambulate independently with or without technical aids
* Barthel Index ≥ 60
* Pre-frailty (1-2 criteria) or Frailty according to the Frailty Phenotype by Fried et al
* Risk of falling according to following criteria:

  * Gait disorders captured through physical performance measures (Time Up and Go Test ≥ 20 s and/or Gait Speed ≥0,8 m/s
  * ≥2 self-reported falls in the previous year
  * ≥1 self-reported falls requiring medical assistance
* Relative/caregiver willingness to supervise the exercise/cognitive stimulation sessions
* Capability and willingness to provide informed consent

Exclusion Criteria:

* Unwillingness to either complete the study requirements or to be randomized into the control or the intervention group
* Life expectancy ≤ 3 months
* Terminal illness
* No possibility of follow-up
* Institutionalization or awaiting institutionalization
* Major cognitive impairment DSM-V moderate or severe (CDR 2-3 /GDS 5-7)
* No ability to read and write
* Severe visual and hearing deficit
* Any contraindications for physical exercise or testing procedures, including but not limited to:

  * myocardial infarction in the past 3 months
  * unstable angina pectoris
  * uncontrolled arrhythmia
  * unstable cardiovascular disease or other unstable medical condition
  * uncontrolled arterial hypertension
  * recent pulmonary thromboembolism
  * upper or lower extremity fracture in the past 3 months

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
One year falls rate | during one year
  Fall: an unexpected event in which the participants come to rest on the ground, floor, or lower level.Subjects will be contacted by phone in a monthly basis after completing the 3-months lasting intervention and inform the research team about the incidence of falls.
One year fall-related hospitalizations | during one year
  Number of fall-related hospitalizations
One year fall-related fracture | during one year
  Number of fall-related fracture (radiologically confirmed)
One year fall-related death | during one year
  Number of fall-related death

SECONDARY OUTCOMES:
Barthel | At baseline, 6-week, 12-week and 24-week and 1-year.
  Barthel Index changes from baseline to 6-week, 12-week and 24-week and 1-year
Garvan Fracture Risk | At baseline and 12-week
  Changes from baseline to 12-week The Fracture Risk Calculator was developed using data collected in the internationally renowned Dubbo Osteoporosis Epidemiology Study conducted by the Bone and Mineral Research Program of Sydney's Garvan Institute of Medical Research. It estimates the 5-year and 10-year risk of hip and any fracture based on information on sex, age, number of fractures since the age of 50, the rate of falling and the bone mineral density.
Handgrip Strength in both hands | At baseline, 6-week, 12-week
  Changes from baseline to 6-week and 12-week.Handgrip strength will be measured by using a dynamometer (JAMAR) in both dominant and non-dominant hand. Best performance of two trials will be registered.
4-metre gait velocity test (GVT) | At baseline, 6 week and 3 months.
  Changes from baseline to 6 week and 3 months.Gait ability will be assessed using the 6-metre gait velocity test (GVT). Starting and ending limits will be marked on the floor with tapelines for a total distance of 8 meters. Participants will be instructed to walk in their self-selected usual pace for two attempts. The best result of both trials will be registered. The first and last metre, considered the warm-up and deceleration phases, respectively, will not be included in calculations of the gait assessment. Higher scores ( > 1.0 m/s) indicates better functional capacity and lower scores (< 0.8 m/s) scores worse functional capacity.
Short Physical Performance Battery (SPPB) | At baseline,1 and 3 months.
  Changes from baseline to 1 and 3 months. The functional capacity of patients will be evaluated by the Short Physical Performance Battery (SPPB) which evaluates, balance, gait ability, and leg strength using a single tool. The total score ranges from 0 (worst) to 12 points (best). The SPPB test has been shown to be a valid instrument for screening frailty and predicting disability, institutionalization, and mortality. A total score of less than 10 indicates frailty and a high risk of disability and falls. A one-point change in the score has clinical relevance
Fried's Frailty Phenotype (FP) | At baseline and 3 months
  Changes from baseline to 3 months. The Fried's Frailty Phenotype (FP) consists of five items: weight loss, exhaustion, strength, physical activity and gait speed. For grip strength, 3-m GS and Physical Activity Scale for the Elderly (PASE) scores. Subjects are classified as robust if not meeting any criteria, pre-frail if they met 1-2 of the criteria and frail if ≥3 were present.
SARC-F (Screening of Sarcopenia Among Older Adults) | At baseline,1 and 3 months.
  Changes from baseline to 1 and 3 months. The SARC-F is a screening scale to ascertain the risk of sarcopenia (the presence of age-associated low muscle mass and function). It is composed of 5 items related to the presence of difficulty in loading weights, walking, standing-up from a chair, climbing stairs and the number of falls in the previous year. A score greater than 4 is indicative of the presence of sarcopenia.
Musculoskeletal echography | At baseline, 6 weeks and 3 months
  Changes from baseline to 6-week and 3 months. Muscle thickness and quality will be assessed through musculoskeletal echography, a non-intrusive imaging method. Muscle thickness and quality (infiltration of non-contractile tissue) will be measured in the rectus femoris (region from sub-cutaneous tissue to the bone surface).
MOCA (Montreal Cognitive Assessment) test | At baseline, 6 weeks and 3 months
  Changes from baseline to 6-week and 3 months. cognitive function will be measured with MOCA ( Montreal Cognitive Assessment Test) in case of mild cognitive decline. The MOCA is a validated test in Spanish It ranges from 0 ( worse score ) to 30 (best score). A score less than 26 indicates suggest mild cognitive decline
Trail Making Test part A ( TMT-A) | At baseline, 6 weeks and 3 months
  Changes from baseline to 6-week and 3 months. Executive function will be assessed with the Trail Making Test part A. Results for TMT A are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.Average will be consider 29 seconds, Deficient > 78 seconds and Rule of Thumb most 90 seconds
Falls-related psychological consequences | At baseline, 12 week, 24 week and 1 year.
  Changes from baseline, 12-week visit; and 24-week and 1-year. Fear of falling will be evaluated through three questions: ''Are you afraid of falling?'', ''Do you limit any house-hold activities because you are frightened you may fall?'', ''Do you limit any outside activities because you are frightened you may fall?''.
  FES-I was developed as part of the Prevention of Falls Network Europe (ProFaNE) project from 2003 to 2006, following an intensive review of fear of falling, self-efficacy and balance confidence questionnaires. It ascertains the impact that fear of falling has on 16 activities of daily living. Scores range from 16 to 64 and classify the fear of falling as low (16-19), moderate (20-27) and high (28-64) concern.
1-Repetition Maximum (RM) Maximal dynamic strength test | At baseline, 6 weeks and 3 months
  Changes from baseline to 6-week and 3 months. Maximal dynamic strength will be assessed using the 1Repetition Maximum (RM) test in the bilateral leg press exercise using exercise machines (Exercycle, S.L., BH Group, Vitoria, Spain). In the first assessment, the subjects will warm up with specific movements for the exercise test. Each subject's maximal load will be determined in no more than five attempts, with a 3-min recovery period between attempts
Repetitions at maximal velocity at intensities of 50% of 1RM test | At baseline, 6 weeks and 3 months
  Changes from baseline to 6-week and 3 months. Participants will perform ten repetitions at maximal velocity at intensities of 50% of 1RM to determine the maximum power (w) and the loss of power during the ten repetitions in the leg press exercise. Higher values indicate better functional capacity
Geriatric Depression Scale (GDS) Yesavage abbreviated scale | At baseline, 6 weeks and 3 months
  Changes from baseline to 6-week and 3 months. Depression will be assessed wit the GDS Yesavage abbreviated scale of 15 items. Is is ranged between 0 ( best value) to 15 ( worse value). Scores between 0-5 indicates normality, 5-9 minor depression and scores over 9 indicates mayor depression
Mortality | At baseline, 6 weeks and 3 months
  Mortality will be assessed with a clinical questionnaire during follow up
Admissions to the hospital | At baseline, 6 weeks and 3 months
  New admissions to the hospital will be assessed with a clinical questionnaire during follow up
Incidence of institutionalization to nursing homes | At baseline, 6 weeks and 3 months
  New institutionalizations to nursing homes will be assessed with clinical questionary during follow up
Visit to emergency room | At baseline, 6 weeks and 3 months
  Visits to emergency room will be assessed with a clinical questionnaire during follow up
Number of total Drugs | At baseline and 3 months
  Number of drugs during follow up will be assessed with a clinical questionnaire
Presence of 5 or more drugs ( Polypharmacy ) registration | At baseline and 3 months
  Registration of the presence of 5 or more drugs( Polypharmacy ) during follow -up will be done with a clinical questionnaire
Psychotropic and hypotensive drugs registration | At baseline and 3 months
  Registration of the presence of psychotropic and hypotensive drugs during follow -up will be done with a clinical questionnaire
Drug Burden Index | At baseline, 3, 6, 9 and 12 months
  It is a pharmacological measure of an individual's exposure to medications with anticholinergic and sedative effects. DBI is calculated for an individual by summing the burdens from every anticholinergic or sedative medicine they take regularly. A calculator available in https://www.anticholinergicscales.es/ will be used.
Dual task gait ( arithmetic) 6 m velocity test | At baseline, week 6 and 3 months
  The dual-task paradigm will be used in the 6-m habitual GVT. Two trials will be conducted (best record will be taking in account) During the arithmetic dual-task condition (arithmetic GVT), we will assess gait velocity while participants are counting backward aloud from 100 by ones
Dual task gait (verbal) 6 m velocity test | At baseline, 6-week and 3 months
  The dual-task paradigm will be used in the 6-m habitual GVT. Two trials will be conducted(best record will be taking in account)During the verbal dual-task condition (verbal GVT), we will assess gait velocity while participants are naming animals by loud
EuroQol-5D (EQ-5D) Quality of life assessment test | At baseline and 3 months
  Quality of life will be assessed with an international validated scale EuroQol-5D (EQ-5D). Its composed by. It asses health status (mobility, personal care, basic and instrumental daily living activities , pain and ansiety/depression) ranged from 0 ( worst health status) to 100 ( best health status )
- Registration of other geriatric syndromes (visual and hear impairment, urinary and fecal incontinence, delirium , dysphagia, constipation , pressure ulcers ) | At baseline and 3 months
  Presence of other geriatric syndromes ( visual and hear impairment, urinary and fecal incontinence, delirium , dysphagia, constipation , pressure ulcers ) will be assessed with a clinical questionnaire

OTHER OUTCOMES:
Mini- Nutritional Assessment (MNA) | At baseline
  The MNA® in the short form (MNA-SF) is a validated nutrition screening and assessment tool that can identify geriatric patients age 65 and above who are malnourished or at risk of malnutrition. Is is ranged from 0 to 14. 12-14 points indicates normal nutritional status : 8-11 points: At risk of malnutrition 0-7 points: Malnourished
Cumulative Illness Rating Scale for Geriatrics (CIRS-G) | At baseline
  This scoring system measures the chronic medical illness ("morbidity") burden while taking into consideration the severity of chronic diseases in 14 items representing individual body systems. The general rules for severity rating are:
  0→No problem affecting that system.
  1. Current mild problem or past significant problem.
  2. Moderate disability or morbidity and/or requires first line therapy.
  3. Severe problem and/or constant and significant disability and/or hard to control chronic problems.
  4. Extremely severe problem and/or immediate treatment required and/or organ failure and/or severe functional impairment.
  The cumulative final score can vary theoretically vary from 0 to 56 (although a very high score is impossible).
Gait regularity analysis with an inertial sensor unit | At baseline, 6-week and3 months
  During functional tasks (such as balance, gait and rising form a chair ) and cognitive evaluations (dual tasking), an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Gait regularity analysis will be performed
Gait cadence analysis with an inertial sensor unit | At baseline, 6-week and3 months
  During functional tasks (such as balance, gait and rising form a chair ) and cognitive evaluations (dual tasking), an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Gait cadence analysis will be performed
Gait variability analysis with an inertial sensor unit | At baseline, 6-week and3 months
  During functional tasks (such as balance, gait and rising form a chair ) and cognitive evaluations (dual tasking), an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Gait variability analysis will be performed
Gait symmetry analysis with an inertial sensor unit - Gait symmetry analysis with an inertial sensor unit | At baseline, 6-week and3 months
  During functional tasks (such as balance, gait and rising form a chair ) and cognitive evaluations (dual tasking), an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Gait symmetry analysis will be performed
Five Times Sit to Stand peak power analysis test with an inertial sensor unit | At baseline, 6-week and3 months
  During functional Five Times to Stand Test an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Peak power analysis will be performed
Five Times Sit to Stand impulse analysis test with an inertial sensor unit | At baseline, 6-week and3 months
  During functional Five Times to Stand Test an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Impulse analysis will be performed
Five Times Sit to Stand orientation analysis test with an inertial sensor unit | At baseline, 6-week and3 months
  During functional Five Times to Stand Test an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Orientation analysis will be performed
Balance power spectrum analysis test with an inertial sensor unit | At baseline, 6-week and3 months
  During functional balance assessment an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Power spectrum analysis will be performed
Balance area analysis test with an inertial sensor unit | At baseline, 6-week and3 months
  During functional balance assessment an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Balance area analysis will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Casas Herrero, MD PhD, Principal Investigator — Fundación Miguel Servet - Navarrabiomed
Locations (1):
- Complejo Hospitalario de Navarra. Department of Geriatrics, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Sanchez-Sanchez JL, Udina C, Medina-Rincon A, Esbri-Victor M, Bartolome-Martin I, Moral-Cuesta D, Marin-Epelde I, Ramon-Espinoza F, Latorre MS, Idoate F, Goni-Sarries A, Martinez-Martinez B, Bonet RE, Librero J, Casas-Herrero A. Effect of a multicomponent exercise program and cognitive stimulation (VIVIFRAIL-COGN) on falls in frail community older persons with high risk of falls: study protocol for a randomized multicenter control trial. BMC Geriatr. 2022 Jul 23;22(1):612. doi: 10.1186/s12877-022-03214-0. PMID 35870875